CLINICAL TRIAL: NCT01958840
Title: Evaluating Behavioral Activation Efficacy in Depressed Spanish-Speaking Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Joe Smith, Director - HRPP (A. Collado is no longer at UMD), University of Maryland, College Park
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1F31MH098512-01A1 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Depression
Keywords: Behavioral; Activation; Treatment
MeSH Terms: conditions — Depression; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Activation Treatment for Depression (Experimental): Behavioral Activation Condition - 10 sessions
  Interventions: Behavioral: Behavioral Activation for Depression Treatment
- Supportive Counseling (Active Comparator): Supportive Counseling Condition - 10 sessions
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Behavioral Activation for Depression Treatment
  Arms: Behavioral Activation Treatment for Depression
Behavioral: Supportive Counseling
  Arms: Supportive Counseling

SUMMARY:
Following a small, open-label pilot study that yielded very promising results of BATD, the current study will consist of a larger, randomized control trial (n=60) that will compare BATD to Supportive Counseling in outcomes of depression, contact with positive reinforcement in the environment, treatment satisfaction, therapeutic alliance, and perceived stigma. In addition, participants' adherence rates to each of the therapies and their maintenance of clinical gains at a 1-month follow-up, will be examined.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is highly prevalent and widely-impairing across racial and ethnic groups. Higher rates of MDD have been observed among Latinos with limited English-language proficiency relative to the general population. Although MDD is a highly treatable condition, barriers to treatment access and delivery have been implicated in precluding this group from utilizing and receiving mental health services. Fortunately, Latinos tend to endorse positive attitudes toward psychosocial treatments for depression by applying the valued belief of "poner de su parte" or being able to do their part in one's recovery, a concept that is highly consistent with the framework of behavioral treatments for depression.

The Behavioral Activation Treatment for Depression (BATD), based on reinforcement theory, may be well-equipped to address disparities associated with higher depression prevalence rates and receipt of care among Latinos with limited English-language proficiency. Following a small, open-label pilot study that yielded very promising results of BATD, the current study will consist of a larger, randomized control trial (N = 60) that will compare BATD to Supportive Counseling in outcomes of depression, activity level, and contact with positive reinforcement in the environment.

Initial eligibility will be determined via a telephone screener, which will include questions from the Mood Disorders, Substance Use and Dependence, and Psychotic Disorders modules of the Structured Clinical Interview for DSM-IV-TR (SCID-IV; First, Spitzer, Gibbon & Williams, 2002).

Inclusion criteria consist of the following: 1) be a minimum of 18 years of age, 2) be of Latino descent, 3) report limited English language proficiency, 4) meet current MDD criteria, 5) have completed the 4th grade or higher either in their country of origin or in the US, 6) not have current substance abuse or dependence, 7) have no Bipolar or Psychotic Disorders, and 9) not be currently receiving psychotherapy, and 10) if currently taking antidepressants, demonstrate pharmacological stability as indicated by 3 or more consecutive months of use. Excluded individuals will be referred to mental health resources within the community.

ELIGIBILITY:
Inclusion Criteria:

* be a minimum of 18 years of age
* be of Latino descent
* report limited English language proficiency
* meet current MDD criteria
* have completed the 4th grade or higher either in their country of origin or in the US
* not have current substance abuse or dependence
* have no Bipolar or Psychotic Disorders
* not be currently receiving psychotherapy
* if currently taking antidepressants, demonstrate pharmacological stability as indicated by 3 or more consecutive months of use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory- II | Assessed at every session and at the 1-month follow-up

SECONDARY OUTCOMES:
Behavioral Activation for Depression Scale | Administered at each session and at the 1-month follow-up

OTHER OUTCOMES:
Reward Probability Index | Administered at each session and at the 1-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland- College Park, College Park, Maryland, United States

REFERENCES:
- [Derived] Collado A, Long KE, MacPherson L, Lejuez CW. The efficacy of a behavioral activation intervention among depressed US Latinos with limited English language proficiency: study protocol for a randomized controlled trial. Trials. 2014 Jun 18;15:231. doi: 10.1186/1745-6215-15-231. PMID 24938081